CLINICAL TRIAL: NCT06121908
Title: Role of Blood Lactate Level in Prediction of Outcome of Cirrhotic Patients at The Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hania Atef Mohamed Abdellatif, Resident of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: Lactate in Cirrhotic Patients
Record Dates: First submitted 2023-10-20; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Liver Cirrhosis
Keywords: Lactate
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Determine in-hospital and 28-days mortality rates of critically-ill cirrhotic patients admitted to ICU
2. Evaluate the role of (blood lactate level, lactate/albumin ratio, lactate/bilirubin index and MELD-lactate score) in prediction of mortality compared to other non- lactate containing scores.
3. Study predictors of in-hospital and 28-mortality in these patients.

DETAILED DESCRIPTION:
Liver cirrhosis is a major health problem, which causes high mortality and economic burden worldwide. A large number of liver cirrhosis patients are prone to acute decompensation with organ failure, thus leading them to be admitted to intensive care unit (ICU).

Though liver cirrhosis patients have improved outcomes in ICU over the past decade, the prognosis for those patients remains poor, with in-hospital mortality. Assessment of prognosis, especially in patients with cirrhosis at the ICU, is of importance in order to guide therapeutic measures and improve their outcome.

Many prognostic scores are used to help predicting complications, expected survival and estimate the risk of various medical interventions in these patients as CTP, MELD, CLIF-C OF, CLIF-C AD and CLIF-C ACLF scores. Although these models are non-invasive, they have certain deficiencies as they don't consider other conditions that are associated with poor prognosis as poor tissue perfusion in critically-ill cirrhotic patients.

Lactate is a marker of metabolic changes resulting from tissue hypoxia or stress caused by the release of adrenaline. It was used to improve the prediction of short-term mortality of critically ill patients at ICU. Little is known about role of blood lactate in prediction of prognosis of critically ill Egyptian cirrhotic patients at ICU. Therefore, the investigators will conduct their study to shed some light on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients who are at least 18 years old at their first ICU admission in Al-Rajhy University Hospital (according to the established admission policy) and stay more than 24 h will be included.

Exclusion Criteria:

* 1) Patients admitted for liver transplantation.
* 2) Patients whose blood lactate data is lost at 24 hours from ICU admission.
* 3) Patients taking drugs that increase level of serum lactate as metformin , acetaminophen, linezolid, epinephrine, beta2 agonists, propofol, nucleoside reverse transcriptase inhibitors (NRTIs) as lamivudine and abacavir , and theophylline

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients who are at least 18 years old at their first ICU admission in Al-Rajhy University Hospital (according to the established admission policy) and stay more than 24 h will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To determine the hospital and 28-days mortality rates in critically-ill cirrhotic patients admitted to ICU of Al-Rajhy Universty Hospital. | within 28 days of patients' admission to the Intensive Care Unit.
  1) To determine the hospital and 28-days mortality rates in critically-ill cirrhotic patients admitted to the Intensive Care Unit of Al-Rajhy Universty Hospital.
To evaluate the role of blood lactate level in prediction of 28-days mortality in critically-ill cirrhotic patients. | Blood lactate level will be estimated on the first day of Patients' admission to the ICU.
  Blood lactate level (mmol/L)
To evaluate the role of lactate/Albumin ratio in prediction of 28-days mortality in critically-ill cirrhotic patients. | Lactate/Albumin ratio will be calculated on the first day of Patients' admission to the ICU.
  Lactate/Albumin ratio (L/A ratio: albumin in (g/L) compared to lactate (mmol/L)).
To evaluate the role of lactate/bilirubin index in prediction of 28-days mortality in critically-ill cirrhotic patients. | Lactate bilirubin index will be calculated on the first day of Patients' admission to the ICU.
  Lactate bilirubin index ( lactate in mmol/L , bilirubin in umol/l ) : will be calculated as follows : [1000 × lactate (mmol/L) × bilirubin (µmol/L)]/2 (Chen et al., 2021).
To evaluate the role of MELD-Lactate score in prediction of 28-days mortality in critically-ill cirrhotic patients. | MELD-Lactate score will be calculated on the first day of Patients' admission to the ICU.
  MELD-Lactate score: (Moreau et al., 2013) will be calculated as follows: 0.251 + 5.5257 × sqrt (lactate mmol/L ) + 0.338 × MELD (Sarmast et al., 2020).

SECONDARY OUTCOMES:
Correlation between blood lactate level and type and number of organ failure. | Within 28 days of Patients' admission to the Intensive Care Unit.
  Correlation between blood lactate level and type and number of organ failure.
Correlation between blood lactate level and duration of hospital stay. | Within 28 days of Patients' admission to the Intensive Care Unit.
  Correlation between blood lactate level and duration of hospital stay.

REFERENCES:
- [Background] Li X, Gong M, Fu S, Zhang J, Wu S. Establishment of MELD-lactate clearance scoring system in predicting death risk of critically ill cirrhotic patients. BMC Gastroenterol. 2022 Jun 3;22(1):280. doi: 10.1186/s12876-022-02351-5. PMID 35658837
- [Background] Drolz A, Horvatits T, Rutter K, Landahl F, Roedl K, Meersseman P, Wilmer A, Kluwe J, Lohse AW, Kluge S, Trauner M, Fuhrmann V. Lactate Improves Prediction of Short-Term Mortality in Critically Ill Patients With Cirrhosis: A Multinational Study. Hepatology. 2019 Jan;69(1):258-269. doi: 10.1002/hep.30151. Epub 2018 Dec 17. PMID 30070381
- [Background] Moon AM, Singal AG, Tapper EB. Contemporary Epidemiology of Chronic Liver Disease and Cirrhosis. Clin Gastroenterol Hepatol. 2020 Nov;18(12):2650-2666. doi: 10.1016/j.cgh.2019.07.060. Epub 2019 Aug 8. PMID 31401364
- [Background] Saliba F, Ichai P, Levesque E, Samuel D. Cirrhotic patients in the ICU: prognostic markers and outcome. Curr Opin Crit Care. 2013 Apr;19(2):154-60. doi: 10.1097/MCC.0b013e32835f0c17. PMID 23426137
- [Background] Weil D, Levesque E, McPhail M, Cavallazzi R, Theocharidou E, Cholongitas E, Galbois A, Pan HC, Karvellas CJ, Sauneuf B, Robert R, Fichet J, Piton G, Thevenot T, Capellier G, Di Martino V; METAREACIR Group. Prognosis of cirrhotic patients admitted to intensive care unit: a meta-analysis. Ann Intensive Care. 2017 Dec;7(1):33. doi: 10.1186/s13613-017-0249-6. Epub 2017 Mar 21. PMID 28321803
- [Background] Fuhrmann V, Whitehouse T, Wendon J. The ten tips to manage critically ill patients with acute-on-chronic liver failure. Intensive Care Med. 2018 Nov;44(11):1932-1935. doi: 10.1007/s00134-018-5078-z. Epub 2018 Jan 31. No abstract available. PMID 29387913
- [Background] Costa E Silva PP, Codes L, Rios FF, Esteve CP, Valverde Filho MT, Lima DOC, de Almeida Filho GF, Morais MCA, Lima BC, Chagas PBO, Boa-Sorte N, Bittencourt PL. Comparison of General and Liver-Specific Prognostic Scores in Their Ability to Predict Mortality in Cirrhotic Patients Admitted to the Intensive Care Unit. Can J Gastroenterol Hepatol. 2021 Sep 24;2021:9953106. doi: 10.1155/2021/9953106. eCollection 2021. PMID 34608435
- [Background] Sarmast N, Ogola GO, Kouznetsova M, Leise MD, Bahirwani R, Maiwall R, Tapper E, Trotter J, Bajaj JS, Thacker LR, Tandon P, Wong F, Reddy KR, O'Leary JG, Masica A, Modrykamien AM, Kamath PS, Asrani SK. Model for End-Stage Liver Disease-Lactate and Prediction of Inpatient Mortality in Patients With Chronic Liver Disease. Hepatology. 2020 Nov;72(5):1747-1757. doi: 10.1002/hep.31199. PMID 32083761
- [Background] Nie Y, Zhang Y, Liu LX, Zhu X. Serum Lactate Level Predicts Short-Term and Long-Term Mortality of HBV-ACLF Patients: A Prospective Study. Ther Clin Risk Manag. 2020 Sep 10;16:849-860. doi: 10.2147/TCRM.S272463. eCollection 2020. PMID 32982257
- [Background] Zanza C, Facelli V, Romenskaya T, Bottinelli M, Caputo G, Piccioni A, Franceschi F, Saviano A, Ojetti V, Savioli G, Longhitano Y. Lactic Acidosis Related to Pharmacotherapy and Human Diseases. Pharmaceuticals (Basel). 2022 Nov 30;15(12):1496. doi: 10.3390/ph15121496. PMID 36558947
- [Background] Chen Xiao-Fu, Zhao Yuan, Chen Wei-Zhen, et al., Lactate and Bilirubin Index: A New Indicator to Predict Critically Ill Cirrhotic Patients' Prognosis, Canadian Journal of Gastroenterology and Hepatology,vol. 2021, Article ID 6624177, 7 pages,2021.
- [Background] Moreau R, Jalan R, Gines P, Pavesi M, Angeli P, Cordoba J, Durand F, Gustot T, Saliba F, Domenicali M, Gerbes A, Wendon J, Alessandria C, Laleman W, Zeuzem S, Trebicka J, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Acute-on-chronic liver failure is a distinct syndrome that develops in patients with acute decompensation of cirrhosis. Gastroenterology. 2013 Jun;144(7):1426-37, 1437.e1-9. doi: 10.1053/j.gastro.2013.02.042. Epub 2013 Mar 6. PMID 23474284